CLINICAL TRIAL: NCT05777239
Title: Dental Implant Approach for Crestal Sinus Elevation; A Novel Technique. Case Series Study
Brief Title: Dental Implant Approach for Crestal Sinus Elevation; A Novel Technique.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDCE.N4
Record Dates: First submitted 2023-03-03; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Maxillary Sinus; Dental Implant; Maxillary Sinus Lift; Maxillary Sinus Elevation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Implant Approach for Crestal Sinus Elevation (Experimental)
  Interventions: Procedure: Dental Implant Approach for Crestal Sinus Elevation

INTERVENTIONS:
Procedure: Dental Implant Approach for Crestal Sinus Elevation — Crestal Sinus Elevation by elevating the sinus membrane with a blunt ended dental implant approach

SUMMARY:
Vertical bone height reduction after extraction in the posterior maxilla is inevitable and complicates the treatment plan. Crestal sinus elevation, using implants and different grafting procedures are considered some of the proposed treatment protocols. Ever since the introduction of implant dentistry and implant placement in the posterior maxilla has been a dilemma. The choice of the type of bone, anatomical landmarks and reduced remaining bone height are all obstacles faced when placing implants in this area. Vertical bone height reduction occurs post extraction of the maxillary molars and premolars by maxillary sinus pneumatization. Many protocols were suggested to overcome this phenomenon; placing short implants, 2nd premolar occlusion and finally maxillary sinus elevation.

A recent systematic review evaluated osteotomes mediated sinus floor elevation with or without grafting material. It concluded a high long term survival rate in both procedures, however only one comparative study was used in the analysis that involved 12 participants only. Another systematic review assessed the survival of implants placed with lateral versus crestal sinus approach in 4-8 mm ridge height. It concluded that the ability of the less invasive crestal sinus approach to replace one-stage lateral approach, however, only one randomized control trial was presented that involved 4o patients, and were followed-up for 5 years. This emphasizes the gap of knowledge in literature with high quality evidence concerning these approaches.

The purpose of the present study is to evaluate the radiographic vertical gain in bone height as well as the implant stability after implant placement without the use of bone grafts in posterior maxilla following sinus elevation using the crestal implant approach technique.

ELIGIBILITY:
Eligibility criteria:

Inclusion criteria:

1. Patients who have at least one missing posterior maxillary tooth with sound adjacent teeth.
2. Adults above the age of 18.
3. Residual Bone height from 5mm to 7mm under the maxillary sinus assessed in CBCT.
4. Mandibular posterior teeth opposing the tooth to be replaced for occlusion.
5. Good oral hygiene.
6. Patient accepts to provide an informed consent.

Exclusion criteria:

1. Smokers.
2. Pregnant and lactating females.
3. Medically compromised patients.
4. Patients with active infection related at the site of implant/bone graft placement.
5. Patients with untreated active periodontal diseases.
6. Patients with parafunctional habits.
7. Acute or chronic sinusitis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Intrasinus bone formation around implant | 1 year
  CBCT mm
Primary stability | 1 day
  torque measure
Surgical complications | 1 year
  Clinical assessment (Yes/No)
Implant Survival | 1 year
  Clinical assessment (Yes/No)

SECONDARY OUTCOMES:
prosthetic complications | 1 year
  Clinical assessment (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Continuing Education, Cairo, Egypt